CLINICAL TRIAL: NCT02824224
Title: Tamoxifen to Reduce Unscheduled Bleeding in New Users of the Levonorgestrel-releasing Intrauterine System (LNG-IUS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Leon Speroff Professor of Obstetrics & Gynecology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00015881
Record Dates: First submitted 2016-07-02; First posted 2016-07-06 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Menorrhagia; Metrorrhagia; Medicated Intrauterine Devices
Keywords: levonorgestrel; breakthrough bleeding
MeSH Terms: conditions — Menorrhagia; Metrorrhagia | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamoxifen (Experimental): Tamoxifen 10mg tablet by mouth twice daily for 7 days
  Interventions: Drug: Tamoxifen
- Placebo (Placebo Comparator): Placebo tablet (for tamoxifen tablet) by mouth twice daily for 7 days
  Interventions: Drug: Placebo (for Tamoxifen)

INTERVENTIONS:
Drug: Tamoxifen — 10mg PO (by mouth) twice daily for 7 days starting on day 21 after IUD insertion for one course
  Other Names: Nolvadex
  Arms: Tamoxifen
Drug: Placebo (for Tamoxifen) — Sugar pill manufactured to mimic the tamoxifen 10mg tablet
  Arms: Placebo

SUMMARY:
This study evaluates the ability of tamoxifen to improve frequent or prolonged bleeding in new users of the 52mg levonorgestrel-releasing intrauterine device (IUD). Half of participants will receive a course of tamoxifen three weeks after insertion of the IUD, while the other half of participants will receive a course of placebo.

DETAILED DESCRIPTION:
New users of the LNG IUD will be eligible. Subjects will be randomized to receive tamoxifen 10 mg twice daily for 7 days or placebo. Study drug will be started 3 weeks after placement of the IUD. Subjects will maintain a record of daily bleeding and spotting using an electronic text messaging diary.

ELIGIBILITY:
Inclusion Criteria:

* initiating use of 52mg levonorgestrel-releasing IUD for contraceptive purposes
* access to reliable cell phone
* willing to receive and respond to daily text or email message to assess bleeding

Exclusion Criteria:

* using IUD for indication other than contraception
* postpartum within 6 months, pregnant, or breastfeeding
* removal and replacement of IUD
* undiagnosed abnormal uterine bleeding prior to placement of IUD
* bleeding dyscrasia
* anti-coagulation use
* active cervicitis
* allergy to tamoxifen
* history of venous thromboembolism
* personal history of breast or uterine malignancy
* use of medication contraindicated with use of tamoxifen (coumadin, letrozole, bromocriptine, rifampicin, aminoglutethimide, phenobarbital)

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan A Cohen, MD, MPH, Study Director — Oregon Health and Science University
Locations (1):
- OHSU Center For Women's Health, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen MA, Simmons KB, Edelman AB, Jensen JT. Tamoxifen for the prevention of unscheduled bleeding in new users of the levonorgestrel 52-mg intrauterine system: a randomized controlled trial. Contraception. 2019 Nov;100(5):391-396. doi: 10.1016/j.contraception.2019.06.009. Epub 2019 Jun 18. PMID 31226322

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n=5) from participation after signing informed consent form. Discontinued IUD (n=1) Declined to participate (n=2) Non-compliant with diaries (n=2)
Period: Overall Study
Arm/Group | Tamoxifen | Placebo
Started | 19 | 18
Completed | 17 | 17
Not Completed | 2 | 1
Not completed — Discontinued, IUS expulsion | 0 | 1
Not completed — Did not show up for allocation visit | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (7.6) | 28.8 (6.1) | 29.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 17 | 13 | 30
  Other | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding and Spotting Days
Description: Mean number of bleeding and spotting days in the tamoxifen group compared to the mean number of bleeding and spotting days in the placebo group
Time Frame: 30 days after initiation of study drug
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 17 | 17
days | 16.8 (9.0) | 12.0 (5.0)

2. Secondary Outcome: Bleeding Pattern Satisfaction
Description: 0-100 mm Visual Analog Scale (VAS) measurement of satisfaction with bleeding pattern. 0 mm = not at all satisfied, 100 mm = very satisfied.
Time Frame: 30 days after initiation of study drug
Population: Only 30 women completed the side effect, satisfaction and acceptability survey (n=15 placebo and n=15 tamoxifen).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 50.7 (28.6) | 58.6 (31.8)

3. Secondary Outcome: IUD Satisfaction
Description: 0-100 mm Visual Analog Scale (VAS) measurement of satisfaction with IUD (intrauterine device). 0 mm = not at all satisfied, 100 mm = very satisfied.
Time Frame: 30 days after initiation of study drug
Population: Only 30 women completed the side effect, satisfaction and acceptability survey (n=15 placebo and n=15 tamoxifen).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 82.7 (22.0) | 75.3 (21.3)

4. Secondary Outcome: Adverse Events
Description: Descriptive reporting of adverse events for each arm
Time Frame: 30 days after initiation of study drug
Population: Adverse event information is reported in "Adverse Event" section of record summary.
Measure: Number; unit: Events
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 17 | 17
Events | 12 | 15

5. Other Pre Specified Outcome: Total Number of Bleeding/Spotting Episodes
Time Frame: 60 days after initiation of study drug
Population: Study ended up only collecting 30-day follow up data
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Number of Prolonged Bleeding Episodes (>8 Days)
Time Frame: 60 days after initiation of study drug
Population: Study ended up only collecting 30-day follow up data
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Longest Bleed-free Interval
Time Frame: 60 days after initiation of study drug
Population: Study ended up only collecting 30-day follow up data
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after initiating study medication.
Arm/Group | Tamoxifen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 12/17 | 15/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen (N=17) | Placebo (N=17)
Hot flashes (General disorders) | 1 | 1
Mood changes (General disorders) | 2 | 5
Headache (General disorders) | 6 | 5
Nausea (General disorders) | 1 | 3
Weight loss (General disorders) | 1 | 0
Fluid retention (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT02824224/Prot_SAP_000.pdf